CLINICAL TRIAL: NCT00046969
Title: Management Of Anemia Under RadioChemotherapy (MARCH): An Open, Randomized Multicenter Study Of The Effect Of NeoRecormon On Treatment Outcome In Patients With Advanced Cervical Cancer Stage IIB -IVA Treated With Primary Simultaneous Radiochemotherapy (Radiotherapy Plus Cisplatin)
Brief Title: Epoetin Beta in Treating Anemia in Patients With Cervical Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AGO Study Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: AGOSG-OVAR-MO16375-MARCH; CDR0000257189 (Registry Identifier: PDQ (Physician Data Query)); EU-20217; ROCHE-MO16375; ROCHE-RO2053859
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2007-03

CONDITIONS: Anemia; Cervical Cancer
Keywords: anemia; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer; cervical adenosquamous cell carcinoma; cervical squamous cell carcinoma; cervical adenocarcinoma
MeSH Terms: conditions — Anemia; Uterine Cervical Neoplasms | interventions — epoetin beta; Cisplatin; Brachytherapy; Radiotherapy

INTERVENTIONS:
Biological: epoetin beta
Drug: cisplatin
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Epoetin beta may stimulate red blood cell production to prevent or control anemia in patients treated with chemotherapy and radiation therapy.

PURPOSE: Randomized phase IV trial to determine the effectiveness of epoetin beta in treating anemia in patients who are receiving cisplatin and radiation therapy for stage IIB, stage III, or stage IVA cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effectiveness of epoetin beta vs standard care for anemia management, in terms of increased hemoglobin levels and the correlation with reduced relapse/treatment failure rate, in patients with stage IIB, III, or IVA cervical cancer treated with cisplatin and radiotherapy.
* Compare the safety of these regimens in these patients.
* Compare the relapse-free and overall survival of patients treated with these regimens.
* Compare the frequency and localization of relapses and metastases in patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.
* Compare the type, frequency, and degree of adverse events in patients treated with these regimens.
* Compare the overall response rate in patients treated with these regimens.

OUTLINE: This is a randomized, open-label, parallel-group, multicenter study. Patients are stratified according to country, disease stage, and brachytherapy technique. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radiotherapy 5 days a week for 6 weeks. Patients also undergo high-dose rate, low-dose rate, or boost brachytherapy. Patients receive cisplatin IV beginning on day 1 of radiotherapy and continuing weekly for 6 weeks. Patients also receive epoetin beta subcutaneously 3 times a week beginning 2 weeks before radiotherapy and continuing for 8 weeks.
* Arm II: Patients undergo radiotherapy and brachytherapy and receive cisplatin as in arm I.

Quality of life is assessed at baseline, after the last treatment, and at 3 months.

Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 80-450 patients will be accrued for this study within 4-22.5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IIB, III, or IVA cervical cancer

  * No chorion carcinoma or neuroendocrine small cell carcinoma
  * Previously untreated disease
* Must be scheduled to undergo radiotherapy and receive cisplatin as primary therapy
* Hemoglobin 8.0-13.0 g/dL
* No relevant acute bleeding within the past 3 months, including anemia caused by gross bleeding from tumor
* No distant metastasis
* No positive para-aortic lymph nodes

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* WHO 0-2

Life expectancy

* At least 3 months

Hematopoietic

* See Disease Characteristics
* WBC greater than 3,000/mm3
* Platelet count greater than 100,000/mm3
* No hemolytic anemia
* No transferrin saturation less than 20% that cannot be treated with IV iron
* No hemoglobinopathies (i.e., sickle cell disease or thalassemia of all types)

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Transaminases no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal

* Creatinine clearance greater than 60 mL/min

Cardiovascular

* No chronic heart failure
* No New York Heart Association class II-IV heart disease
* No uncontrolled arterial hypertension (systolic blood pressure at least 170 mmHg, diastolic blood pressure at least 100 mmHg)
* No prior deep vein thrombosis
* No thrombocytosis

Other

* No vitamin B12 deficiency
* No folic acid deficiency
* No newly diagnosed (unstable) epilepsy
* No acute infection
* No other malignancy within the past 5 years except basal cell carcinoma in situ
* No known peripheral neuropathy or moto-sensory neurotoxicity grade 2 or greater
* No impaired hearing grade 2 or greater
* No hypersensitivity to benzyl alcohol, benzoic acid, benzalkonium chloride, or any excipients of cisplatin preparations
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 months since prior epoetins or related compounds

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy for cervical cancer

Surgery

* Not specified

Other

* At least 30 days since prior investigational drugs
* No prior systemic antineoplastic therapy for cervical cancer
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2002-07; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Number of treatment failures within 6 months after beginning radiochemotherapy (RCT) (stage I)
Overall survival after RCT (stage II)

SECONDARY OUTCOMES:
Progression/relapse-free survival
Overall response rate to RCT
Overall survival after RCT (stage I)
Frequency and localization of relapses and/or metastases
Change in hemoglobin from baseline during therapy
Quality of life as assessed by the Functional Assessment of Cancer Therapy-Anemia
Type, frequency, and degree of adverse events
Safety
Vital signs
Number of treatment failures within 6 months after beginning RCT (stage II)

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Koelbl, MD, Study Chair — Martin-Luther-Universität Halle-Wittenberg
Locations (1):
- Martin Luther Universitaet, Halle, Germany